CLINICAL TRIAL: NCT03355846
Title: Pain and Bleeding in Subjects With Acute Anal Fissure: Comparative Evaluation of Three Treatments
Acronym: PBSAAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Massimo Chiaretti, Reasercher, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URomLS-2017-1
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2017-11

CONDITIONS: Acute Anal Fissure
Keywords: Anal Fissure; local therapy; pain; defecation; bleeding
MeSH Terms: conditions — Fissure in Ano; Pain; Hemorrhage | interventions — Centella asiatica extract

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- AAF treated with Centella® Complex (Experimental): Centella® Complex 1 cps 60 mg per os
  Interventions: Drug: Centella
- AAF treated with Proctocella® cream (Experimental): Proctocella® Complex cream to be applied in anal area and anal canal
  Interventions: Drug: Proctocella
- AAF treated with Flavonil® cps (Experimental): Flavonil® 1 cps 300 mg per os
  Interventions: Drug: Flavonil® cps
- AAF treated with Flavonil® Cream (Experimental): Flavonil® Cream Cream to be applied in anal region and anal canal
  Interventions: Drug: Flavonil® Cream
- AAF treated with Rectalgan Mousse (Experimental): Rectalgan Mousse cleansing cleanser for anal and perineal region
  Interventions: Drug: Rectalgan Mousse

INTERVENTIONS:
Drug: Centella — after meals twice a day for 15 days
  Arms: AAF treated with Centella® Complex
Drug: Proctocella — after hygiene treatment for 4 weeks;
  Arms: AAF treated with Proctocella® cream
Drug: Flavonil® cps — after meals twice a day for 15 days
  Arms: AAF treated with Flavonil® cps
Drug: Flavonil® Cream — treatment for 4 weeks;
  .
  Arms: AAF treated with Flavonil® Cream
Drug: Rectalgan Mousse — for 4 weeks
  Arms: AAF treated with Rectalgan Mousse

SUMMARY:
Starting from the observation that acute anal fissure (AAF) in 6-8 weeks can heal spontaneously and that some of the commonly used commercial products in clinical practice would seem to be useful, the rationale of the comparative study is to try to identify, in compliance with the protocol of Helsinki (2013), the most effective short-term treatment for the disappearance of pain in defecation and cessation of bleeding, shortening the duration of the healing process and favoring the patient's rapid return to his / her activity, respect for patient safety.

DETAILED DESCRIPTION:
Starting from the observation that anal fissure in 6-8 weeks can heal spontaneously and that some of the commonly used commercial products in clinical practice would seem to be useful, the rationale of the comparative study is to try to identify, in compliance with the protocol of Helsinki (2013), the most effective short-term treatment for the disappearance of pain in defecation and cessation of bleeding, shortening the duration of the healing process and favoring the patient's rapid return to his / her activity, respect for patient safety.

The comparative study will be conducted by comparing the following products:

* Centella® Complex 1 cps 60 mg per os after meals twice a day for 15 days;
* Proctocella® Complex cream to be applied in anal area and anal canal after hygiene treatment for 4 weeks;
* Flavonil® 1 cps 300 mg per os after meals twice a day for 15 days;
* Flavonil® Cream Cream to be applied in anal region and anal canal after hygiene treatment for 4 weeks;
* Rectalgan Mousse cleansing cleanser for anal and perineal region for 4 weeks.

Our approach attempts to blend, based on the evidence of the most recent scientific literature, the experience of decades of colonproctologic clinical practice that has a predominantly surgical approach, with the clinical evidence of the Science of Nutrition which has a conservative vision in the treatment of ailments and constipation, a predisposing factor in the pathogenesis of anal fissure, in order to obtain healing without surgery. The control group will receive the traditional basic treatment consisting in the application of lubricated anal dilators of increasing gauge according to predetermined pattern, hygiene and diet. The two groups with which they will be compared for the results will receive, in addition to the foregoing (for controls), or Flavonoids (ProtFlav) or Asian Centella Extract (ProtCent), in the form of local mouth and cream tablets to be applied at the perianal level and possibly in the anal canal with gloved finger, containing the same active principles also administered by mouth.

ELIGIBILITY:
Inclusion Criteria:

* Subjects With Acute Anal Fissure
* Collaborative patients able to understand and want;

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
time for the disappearance of pain | 1 month
  time for the disappearance of pain in course of treatment

SECONDARY OUTCOMES:
time for the disappearance of bleeding | 1 month
  time for the disappearance of bleeding in course of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery "Paride Stefanini", University of Rome "La Sapienza", Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim DW, Chi YS, Son KH, Chang HW, Kim JS, Kang SS, Kim HP. Effects of sophoraflavanone G, a prenylated flavonoid from Sophora flavescens, on cyclooxygenase-2 and in vivo inflammatory response. Arch Pharm Res. 2002 Jun;25(3):329-35. doi: 10.1007/BF02976635. PMID 12135106
- [Background] Basile M, Gidaro S, Pacella M, Biffignandi PM, Gidaro GS. Parenteral troxerutin and carbazochrome combination in the treatment of post-hemorrhoidectomy status: a randomized, double-blind, placebo-controlled, phase IV study. Curr Med Res Opin. 2001;17(4):256-61. PMID 11922398
- [Background] Mullen W, McGinn J, Lean ME, MacLean MR, Gardner P, Duthie GG, Yokota T, Crozier A. Ellagitannins, flavonoids, and other phenolics in red raspberries and their contribution to antioxidant capacity and vasorelaxation properties. J Agric Food Chem. 2002 Aug 28;50(18):5191-6. doi: 10.1021/jf020140n. PMID 12188628
- [Background] Jantet G. Chronic venous insufficiency: worldwide results of the RELIEF study. Reflux assEssment and quaLity of lIfe improvEment with micronized Flavonoids. Angiology. 2002 May-Jun;53(3):245-56. doi: 10.1177/000331970205300301. PMID 12025911
- [Background] Misra MC, Parshad R. Randomized clinical trial of micronized flavonoids in the early control of bleeding from acute internal haemorrhoids. Br J Surg. 2000 Jul;87(7):868-72. doi: 10.1046/j.1365-2168.2000.01448.x. PMID 10931020
- [Result] Chiaretti M, Fegatelli DA, Ceccarelli G, Carru GA, Pappalardo G, Chiaretti AI. Comparison of Flavonoids and Centella asiatica for the treatment of chronic anal fissure. A randomized clinical trial. Ann Ital Chir. 2018;89:330-336. PMID 29844250